CLINICAL TRIAL: NCT03398668
Title: Combined Occipital and Supraorbital Transcutaneous Nerve Stimulation for Treatment of Migraine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Neurolief Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SP301
Record Dates: First submitted 2018-01-08; First posted 2018-01-12 (Actual); Last update posted 2019-03-13 (Actual); Status verified 2019-03

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Relievion device- Treatment stimulation (Active Comparator): Relievion Device- Treatment combined occipital and supraorbital transcutaneous nerve stimulation
  Interventions: Device: Relievion device- Treatment stimulation
- Sham Comparator: Relievion device- Sham Stimulation (Sham Comparator): Relievion Device- Sham combined occipital and supraorbital transcutaneous nerve stimulation
  Interventions: Device: Relievion Device- Sham stimulation

INTERVENTIONS:
Device: Relievion device- Treatment stimulation — 1 Hour self-administered treatment specific occipital and supraorbital transcutaneous nerve stimulation
  Other Names: Neurolief device
  Arms: Relievion device- Treatment stimulation
Device: Relievion Device- Sham stimulation — 1 Hour self-administered sham occipital and supraorbital transcutaneous nerve stimulation
  Other Names: Sham Neurolief device
  Arms: Sham Comparator: Relievion device- Sham Stimulation

SUMMARY:
This study will evaluate the clinical performance and safety of a self administered abortive treatment for migraine headache using combined occipital and supraorbital transcutaneous nerve stimulator (Neurolief device, Relievion™).

ELIGIBILITY:
Inclusion Criteria:

1. Males and females Ages of 18 to 65 years old.
2. History of episodic or chronic migraine with or without aura meeting the diagnostic criteria listed in ICHD (International Classification of Headache Disorders)-III beta (2013) section 1, migraine, with the exception of ''complicated migraine'' (i.e., hemiplegic migraine, basilar-type migraine, ophthalmoplegic migraine, migrainous infarction).
3. Capable to corporate with the study protocol and to sign an informed consent.

Exclusion Criteria:

1. Patients having received Botox treatment in the head region in the prior 4 months.
2. Patients having received supraorbital or occipital nerve blocks in the prior 4 months.
3. History of Medication Overuse Headache.
4. Patients using opioid medication.
5. Allodynia: intolerance to supraorbital and/or occipital neurostimulation that makes the treatment not applicable (the patients will be excluded if they are unable to tolerate the first 10 minutes of neurostimulation).
6. Implanted metal or electrical devices in the head (not including dental implants).
7. Patient having had a previous experience with the Relievion™ device.
8. Patients who have concomitant epilepsy.
9. History of neurosurgical interventions.
10. Patients with implanted neurostimulators, surgical clips (above the shoulder line) or any medical pumps.
11. History of drug abuse or alcoholism.
12. Participation in current clinical study or participated in a clinical study within 3 months prior to this study.
13. Skin lesion or inflammation at the region of the stimulating electrodes.
14. Personality or somatoform disorder.
15. Pregnancy or Lactation.
16. Women with child bearing potential without medically acceptable method of contraception.
17. History of cerebrovascular event.
18. Subjects with recent brain or facial trauma (occurred less than 3 months prior to this study).
19. Patients using Cannabis
20. Patients with head circumference smaller than 51 centimeters or head circumference larger than 60 centimeters.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2018-02-22 (Actual); Primary Completion 2018-12-30 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
Mean change of pain score (measured on a visual analog scale=VAS) at 1 hour compared to baseline | 1 hour
  visual analog scale (VAS) for pain score assessment: 11 point scale 0-no pain, 10-Intolerable pain

SECONDARY OUTCOMES:
Mean change of pain score (measured by VAS) at 2 hours compared to baseline (if rescue therapy was not used). | 2 hours
  visual analog scale (VAS) for pain score assessment: 11 point scale 0-no pain, 10-Intolerable painbaseline (if rescue therapy was not used).
Mean change of pain score (measured by VAS) at 24 hours compared to baseline (if rescue therapy was not used). | 24 hours
  Mean change of pain score (measured by VAS) at 24 hours compared to baseline (if rescue therapy was not used).
Proportion of patients not having required rescue medication within 24 hours | 24 hours
  Proportion of patients not having required rescue medication within 24 hours
Proportion of patients not having required rescue medication at 2 hours compared to baseline. | 2 hours
  Proportion of patients not having required rescue medication at 2 hours
Proportion of patients pain free at 1,2 and 24 hours from baseline (if rescue therapy was not used). | 1, 2, 24 hours
  Proportion of patients pain free at 1,2 and 24 hours from baseline (if rescue therapy was not used).
Proportion of "responders" ("responder" is defined as decrease of at least 50% in VAS pain score from baseline) at 1,2 and 24 hours from baseline (if rescue therapy was not used). | 1, 2, 24 hours
  visual analog scale (VAS) for pain score assessment: 11 point scale 0-no pain, 10-Intolerable pain

OTHER OUTCOMES:
Safety endpoints will consist of recording of adverse events and serious adverse events during the study. Device related adverse events will be evaluated between study groups | 1, 2, 24 hours
  Safety endpoints will consist of recording of adverse events and serious adverse events during the study. Device related adverse events will be evaluated between study groups

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Dr. Oved, Dr., Principal Investigator — Laniado Medical center
Locations (1):
- Laniado Medcial Center, Netanya, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Daniel O, Tepper SJ, Deutsch L, Sharon R. External Concurrent Occipital and Trigeminal Neurostimulation Relieves Migraine Headache: A Prospective, Randomized, Double-Blind, Sham-Controlled Trial. Pain Ther. 2022 Sep;11(3):907-922. doi: 10.1007/s40122-022-00394-w. Epub 2022 Jun 4. PMID 35661128